CLINICAL TRIAL: NCT07024537
Title: Hepatic Arterial Infusion Pump (HAIP) Combined With Fuquinitinib as Late-line Treatment in Patients With Colorectal Cancer Liver Metastases（CRLM）: A Phase 2 Single-Arm Clinical Trial
Brief Title: HAIP Combined With Fuquinitinib as Late-line Treatment in Patients With CRLM：A Phase 2 Single-Arm Clinical Trial
Acronym: HAIP，CRLM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Meng Qiu (Other)
Responsible Party: Sponsor-Investigator, Meng Qiu, Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Approval No. 380, 2024
Record Dates: First submitted 2025-05-26; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A Phase II Single-Arm Clinical Trial (Experimental): All patients received FOLFOXIRI-HAIP chemotherapy and oral fruquintinib. All patients received oral fruquintinib at an initial dose of 4 mg once daily from day 1 to day 21 of each 28-day cycle, and FOLFOXIRI-HAIP chemotherapy with Oxaliplatin 85 mg/m² and Leucovorin 400 mg/m² infused via arterial pump over 2 hours on day 1, Irinotecan 150 mg/m² infused via arterial pump over 90 minutes on day 1,and 5-Fluorouracil 2400 mg/m² infused via arterial pump over 46 hours, repeated biweekly until disease progression, patient's refusal, unacceptable toxic effects, or withdrawal of consent.
  Interventions: Drug: FOLFOXIRI-HAIP+Fuquinitinib

INTERVENTIONS:
Drug: FOLFOXIRI-HAIP+Fuquinitinib — All patients received oral fruquintinib at an initial dose of 4 mg once daily from day 1 to day 21 of each 28-day cycle, and FOLFOXIRI-HAIP chemotherapy with Oxaliplatin 85 mg/m² and Leucovorin 400 mg/m² infused via arterial pump over 2 hours on day 1, Irinotecan 150 mg/m² infused via arterial pump over 90 minutes on day 1,and 5-Fluorouracil 2400 mg/m² infused via arterial pump over 46 hours, repeated biweekly until disease progression, patient's refusal, unacceptable toxic effects, or withdrawal of consent.

SUMMARY:
This study was a phase 2, single-arm, single-center clinical trial in which previously treated patients with unresectable colorectal cancer liver metastases.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the safety and efficacy of hepatic arterial infusion pump chemotherapy combined with fruquintinib in later treatment for colorectal cancer liver metastases. All patients received FOLFOXIRI-HAIP chemotherapy and oral fruquintinib. The primary end point was objective response rate (ORR), and the secondary endpoints were disease control rate (DCR), the liver-specific ORR, overall survival (OS), progression-free survival (PFS), liver-specific PFS, and safety.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years;
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 to 2;
* Prior treatment with chemotherapy based on oxaliplatin, fluorouracil, and irinotecan, with or without EGFR or VEGFR monoclonal antibodies;
* at least one measurable intrahepatic target lesion according to RECIST V1.1 criteria
* normal major organ function

Exclusion Criteria:

* previous treatment with transarterial chemoembolization (TACE) or HAIC;2) prior use of fruquintinib
* presence of other systemic primary malignancies, excluding colorectal cancer
* allergy to the study drug;5) Severe dysfunction of major organs (liver, kidney, heart, or lungs)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate | The best evaluation of clinical efficacy from the time of the first initiation of treatment until the patient's disease progression to change of treatment or death, assessed up to 100 months.
  ORR is defined as the proportion of patients with the best overall response of CR or PR among all participants.

SECONDARY OUTCOMES:
overall progression-free survival (PFS) | From date of the first treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  PFS is defined as the time from the initiation of treatment until disease progression or death.
overall survival (OS) | From date of the first treatment until the date of date of death from any cause,assessed up to 100 months.
  OS is defined as the time from the initiation of treatment until the patient is lost to follow-up or death.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Qiu, Professor, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
First of all, there is a lack of sufficient funds or personnel to anonymize and maintain the data for a long time, such as the original imaging documents, which are difficult to organize compliance. Second, this study was an early exploratory study with small data size and high risk of identification. Finally, summary results are available after publication, and the data will be reassessed 5 years after the end of the study.

REFERENCES:
- [Background] Mayer RJ, Van Cutsem E, Falcone A, Yoshino T, Garcia-Carbonero R, Mizunuma N, Yamazaki K, Shimada Y, Tabernero J, Komatsu Y, Sobrero A, Boucher E, Peeters M, Tran B, Lenz HJ, Zaniboni A, Hochster H, Cleary JM, Prenen H, Benedetti F, Mizuguchi H, Makris L, Ito M, Ohtsu A; RECOURSE Study Group. Randomized trial of TAS-102 for refractory metastatic colorectal cancer. N Engl J Med. 2015 May 14;372(20):1909-19. doi: 10.1056/NEJMoa1414325. PMID 25970050
- [Background] Verheij FS, Kuhlmann KFD, Silliman DR, Soares KC, Kingham TP, Balachandran VP, Drebin JA, Wei AC, Jarnagin WR, Cercek A, Kok NFM, Kemeny NE, D'Angelica MI. Combined Hepatic Arterial Infusion Pump and Systemic Chemotherapy in the Modern Era for Chemotherapy-Naive Patients with Unresectable Colorectal Liver Metastases. Ann Surg Oncol. 2023 Dec;30(13):7950-7959. doi: 10.1245/s10434-023-14073-3. Epub 2023 Aug 28. PMID 37639032
- [Background] Prager GW, Taieb J, Fakih M, Ciardiello F, Van Cutsem E, Elez E, Cruz FM, Wyrwicz L, Stroyakovskiy D, Papai Z, Poureau PG, Liposits G, Cremolini C, Bondarenko I, Modest DP, Benhadji KA, Amellal N, Leger C, Vidot L, Tabernero J; SUNLIGHT Investigators. Trifluridine-Tipiracil and Bevacizumab in Refractory Metastatic Colorectal Cancer. N Engl J Med. 2023 May 4;388(18):1657-1667. doi: 10.1056/NEJMoa2214963. PMID 37133585
- [Background] Li J, Qin S, Xu R, Yau TC, Ma B, Pan H, Xu J, Bai Y, Chi Y, Wang L, Yeh KH, Bi F, Cheng Y, Le AT, Lin JK, Liu T, Ma D, Kappeler C, Kalmus J, Kim TW; CONCUR Investigators. Regorafenib plus best supportive care versus placebo plus best supportive care in Asian patients with previously treated metastatic colorectal cancer (CONCUR): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2015 Jun;16(6):619-29. doi: 10.1016/S1470-2045(15)70156-7. Epub 2015 May 13. PMID 25981818
- [Background] Levi FA, Boige V, Hebbar M, Smith D, Lepere C, Focan C, Karaboue A, Guimbaud R, Carvalho C, Tumolo S, Innominato P, Ajavon Y, Truant S, Castaing D, De Baere T, Kunstlinger F, Bouchahda M, Afshar M, Rougier P, Adam R, Ducreux M; Association Internationale pour Recherche sur Temps Biologique et Chronotherapie (ARTBC International). Conversion to resection of liver metastases from colorectal cancer with hepatic artery infusion of combined chemotherapy and systemic cetuximab in multicenter trial OPTILIV. Ann Oncol. 2016 Feb;27(2):267-74. doi: 10.1093/annonc/mdv548. Epub 2015 Nov 16. PMID 26578731
- [Background] Li J, Qin S, Xu RH, Shen L, Xu J, Bai Y, Yang L, Deng Y, Chen ZD, Zhong H, Pan H, Guo W, Shu Y, Yuan Y, Zhou J, Xu N, Liu T, Ma D, Wu C, Cheng Y, Chen D, Li W, Sun S, Yu Z, Cao P, Chen H, Wang J, Wang S, Wang H, Fan S, Hua Y, Su W. Effect of Fruquintinib vs Placebo on Overall Survival in Patients With Previously Treated Metastatic Colorectal Cancer: The FRESCO Randomized Clinical Trial. JAMA. 2018 Jun 26;319(24):2486-2496. doi: 10.1001/jama.2018.7855. PMID 29946728
- See also: Pubmed Official website — https://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Analytic Code: Statistical analysis — http://www.Rproject.org — The Kaplan-Meier method was used to analyze OS and PFS in the overall population with estimated medians and 95% CIs presented. Survival curves were performed using R software version 4.2.2 (http://www.Rproject.org).

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT07024537/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT07024537/ICF_001.pdf